CLINICAL TRIAL: NCT05255445
Title: Red Blood Cell - IMProving trAnsfusions for Chronically Transfused Recipients (RBC-IMPACT)
Brief Title: Red Blood Cell - IMProving trAnsfusions for Chronically Transfused Recipients
Acronym: RBC-IMPACT
Status: Completed | Type: Observational
Sponsor: Westat (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 75N92019D00032; 75N92019D00033 (Other Grant/Funding Number: National Heart, Lung and Blood Institute); 75N92019D00034 (Other Grant/Funding Number: National Heart, Lung and Blood Institute); 75N92019D00035 (Other Grant/Funding Number: National Heart, Lung and Blood Institute); 75N92019D00036 (Other Grant/Funding Number: National Heart, Lung and Blood Institute); 75N92019D00037 (Other Grant/Funding Number: National Heart, Lung and Blood Institute); 75N92019D00038 (Other Grant/Funding Number: National Heart, Lung and Blood Institute)
Record Dates: First submitted 2022-02-10; First posted 2022-02-24 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease; Thalassemia; Pediatric Cancer
Keywords: Transfusion; Red Blood Cell; Sickle Cell Disease; Thalassemia; Pediatric; Oncology; RBC survival; Genetic; Non-genetic; Observational; Blood donor
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Neoplasms | interventions — Erythrocyte Count; Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens to be stored for future use from enrolled red cell transfusion recipients include whole blood, plasma and serum.
  The study will also retain a sample of packed RBCs from the transfused RBC unit, and a retention tube from the donor of that transfused unit (to be used for extended genotyping but not retained in a long-term biorepository).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Sickle cell disease (SCD): Patients with SCD who are chronically transfused (in the U.S. and Brazil)
  Interventions: Biological: Red Blood Cell (RBC) Transfusion
- Thalassemia: Patients with thalassemia who are chronically transfused in the U.S.
  Interventions: Biological: Red Blood Cell (RBC) Transfusion
- Pediatric Hematology-Oncology: Patients in U.S. with pediatric oncologic diagnoses with hypo-proliferative bone marrow requiring single unit red blood cell transfusion
  Interventions: Biological: Red Blood Cell (RBC) Transfusion
- Blood Donors: Allogenic blood donors in the US (estimated: 10,200) and allogenic blood donors in Brazil (estimated: 2,100) with extended donation genotyping using an investigational hematology array.

INTERVENTIONS:
Biological: Red Blood Cell (RBC) Transfusion — Simple RBC transfusion or partial manual exchange
  Groups: Pediatric Hematology-Oncology; Sickle cell disease (SCD); Thalassemia

SUMMARY:
Red Blood Cell - IMProving trAnsfusions for Chronically Transfused recipients (RBC-IMPACT) is an observational cohort study to assess donor, component, and recipient factors that contribute to RBC efficacy in chronically and episodically transfused patients. The objective of the study is to determine how specific genetic and non-genetic factors in donors and recipients may impact RBC survival after transfusion - in short, what factors on both the donor and recipient side may improve the efficacy of the transfusion.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) and thalassemia are genetic disorders inducing anemia of differing pathophysiology. A primary therapy for preventing certain SCD complications (e.g., stroke) and for thalassemia major is regular red blood cell (RBC) transfusion, coupled with iron chelation to prevent the complications of transfusion-induced iron overload. For patients with pediatric hematology-oncology diagnoses with chemotherapy-induced aplasia, RBC transfusion is also common, but the degree of transfusion-induced iron overload and its implications for these patients is incompletely understood. Because iron-related tissue toxicity is a major cause of morbidity and mortality in regularly transfused patients, developing strategies to minimize iron loading and iron toxicity is a key objective of this proposal (study Aim #2), stemming from the objective to optimize RBC unit characteristics that patients with SCD and thalassemia receive beyond RBC phenotype matching for Rh C, E and K antigens (study Aim #1). The study will enroll patients with SCD, thalassemia or pediatric oncologic diagnoses receiving eligible transfusion at 6 hospital sites in the United States, as well as patients with SCD at 5 hemocenters in Brazil.

ELIGIBILITY:
Inclusion Criteria (Aim #1):

* Well-characterized transfusion-dependent form of SCD or thalassemia (including Hemoglobin E-thalassemia and sickle-beta thalassemia) on chronic simple transfusion therapy or partial manual exchange
* On a regular simple RBC transfusion schedule, including partial manual exchange (i.e., 1-3 units scheduled every 2-6 weeks and on a minimum 6-month chronic transfusion trial; for partial manual exchange, the phlebotomy must be completed before the transfusion is started without a back and forth between rounds of phlebotomy and transfusion)
* Seen at any participating domestic hub hospital (i.e., Columbia University Irving Medical Center/Morgan Stanley Children's Hospital of New York, Weill Cornell Medical Center/Komansky Children's Hospital, Boston Children's Hospital, Froedtert & Medical College of Wisconsin/Children's Wisconsin, University of California San Francisco, Benioff Children's Hospital Oakland) or enrolled in the Brazil REDS-IV-P sickle cell disease cohort and seen at any participating Brazil hemocenter (i.e., Childrens Institute and Adult Clinics at Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HCFMUSP, HEMOAM - Amazonas, HEMOMINAS - Minas Gerais, HEMOPE -Pernambuco, and HEMORIO - Rio de Janeiro)

Exclusion Criteria (Aim #1):

* Institutionalization or imprisonment
* Foster care
* Weight <11 kg

Inclusion criteria (Aim #2):

* Either included in Aim #1 (consented patient with SCD or thalassemia) or patient with pediatric oncologic diagnosis under care in a pediatric hematology/oncology service with anemia due to chemotherapy or primary/secondary hypo-proliferative bone marrow requiring a RBC transfusion (including HSCT)
* [In domestic study only] Age ≤21 years old (many pediatric services include care of patients up to age 21, therefore the protocol will not limit by age but instead on whether they are seen in a pediatric service)
* Planned transfusion of RBC from an aliquot or unit from a single donor
* Seen at any participating domestic hub hospital (i.e., Columbia University Irving Medical Center/Morgan Stanley Children's Hospital of New York, Weill Cornell Medical Center/Komansky Children's Hospital, Boston Children's Hospital, Froedtert & Medical College of Wisconsin/Children's Wisconsin, University of California San Francisco, Benioff Children's Hospital Oakland) or at any REDS-IV-P participating Brazil hemocenter (i.e., Childrens Institute and Adult Clinics at Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HCFMUSP, HEMOAM - Amazonas, HEMOMINAS - Minas Gerais, HEMOPE -Pernambuco, and HEMORIO - Rio de Janeiro).

Exclusion criteria (Aim #2):

* Institutionalization or imprisonment
* Foster care
* Current active auto-immune hemolytic anemia based on positive direct antiglobulin test (DAT) with laboratory evidence of hemolysis and increased transfusion requirement
* [In domestic study only] Microangiopathic hemolytic anemia
* Weight <18 kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All transfused patients with sickle cell disease (in the U.S or Brazil) and thalassemia on simple chronic transfusion (or partial manual exchange transfusion) from hospitals affiliated with REDS-IV-P Domestic hubs or Brazil hemocenters. (Aim #1)
  Chronically transfused patients with sickle cell disease or thalassemia, and patients with pediatric oncology diagnoses with hypo-proliferative bone marrow receiving care at hospitals affiliated with REDS-IV-P Domestic hubs or Brazil hemocenters (for SCD only). (Aim #2).
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A or Hemoglobin Level per day (RBC Survival) | Baseline (immediately pre-) to post-transfusion over 2 years
  Change in hemoglobin A or hemoglobin level per day in between subsequent transfusion episodes, for sickle cell disease and thalassemia cohorts, respectively
Change in Serum Iron Level | Baseline (immediately before) and 2-hours after transfusion
  For all groups participating, change in serum iron measured from immediately prior to 2 hours post-transfusion

SECONDARY OUTCOMES:
Hemoglobin Increment | Baseline (immediately pre-) to post-transfusion, over 2 years
  Hemoglobin increment [defined as Hb/HbA(post-transfusion)visit(i) - Hb/HbA(pre-transfusion)visit(i)] is associated with "RBC survival"
Hemolysis Parameter Increment | Baseline (immediately pre-) to post-transfusion or 2-hours post-transfusion, over 2 years
  Includes serum iron, indirect bilirubin, or plasma free hemoglobin
Hepcidin Level | Baseline (immediately before) to 2 hours after transfusion
  Hepcidin level at time of transfusion is a predictor of change in iron parameters (i.e., transferrin saturation, serum iron) following transfusion
Non-Transferrin-Bound Iron (NTBI) Level | Baseline (immediately before) to 2 hours after transfusion
  NTBI levels in patients with pediatric oncologic diagnoses with aplasia are elevated at baseline and increase following transfusion
Number of Clinical Complications | 2 years
  Increased NTBI, serum iron, or transferrin saturation following transfusion is associated with increased risk of clinical adverse effects (i.e., new infections, SCD complications)

OTHER OUTCOMES:
Rate of Alloimmunization | 2 years
  Rate of new alloantibody formation
4-hydroxynonenal [4-HNE] | 2 years
  Recipient oxidative stress pre-transfusion is associated with "RBC survival"
Type I interferon (i.e., MxA protein assay) and other cytokines (i.e., IL-6, MCP-1, IFNgamma) | 2 years
  Recipient inflammation pre-transfusion is associated with "RBC survival"
Number of Transfusion Reactions | 2 years
  Transfusion reactions are associated with "RBC survival"

CONTACTS AND LOCATIONS:
Overall Officials: Eldad A Hod, MD, Principal Investigator — Columbia University; Brian Custer, PhD, MPH, Principal Investigator — Vitalant Research Institute
Locations (14):
- United States (9):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Vitalant Research Institute, San Francisco, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Weill Cornell Medical Collection (WCMC)/New York Presbyterian Hospital (NYPH), New York, New York
  - Columbia University Irving Medical Center/New York Presbyterian Hospital (NYPH), New York, New York
  - New York Blood Center (NYBC), New York, New York
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
  - Versiti Wisconsin, Inc., Milwaukee, Wisconsin
- Brazil (5):
  - HEMOAM - Amazonas, Manaus, Amazonas
  - HEMOMINAS - Minas Gerais, Belo Horizonte, Minas Gerais
  - HEMOPE - Pernambuco, Recife, Pernambuco
  - HEMORIO - Rio De Janeiro, Rio de Janeiro
  - Childrens Institute and Adult Clinics at Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
De-identified public use datasets will be created and delivered to NHLBI at the end of the study (and end of the REDS-IV-P program) and will be made available indefinitely for future analysis
Supporting Information: Study Protocol, CSR
Time Frame: At the end of the REDS-IV-P program, estimated in March 2026, the public use data sets will be available and will be available indefinitely for future analytic use.
Access Criteria: Public use datasets will be posted to NIH/NHLBI data repository systems.

REFERENCES:
- [Derived] Karafin MS, Kelly S, Chapman KM, Kreuziger LB, Manis JP, Dinardo C, Josephson CD, Stone M, Roubinian NH, Branchford B, Sachais BS, Hailu B, Sabino EC, Hod EA, Custer B; National Heart, Lung, and Blood Institute (NHLBI) Recipient Epidemiology and Donor Evaluation Study-IV-Pediatric (REDS-IV-P). The Red Blood Cell-Improving Transfusions for Chronically Transfused Recipients (RBC-IMPACT) study: protocol description of an international multi-site observational clinical study. Blood Transfus. 2025 Sep-Oct;23(5):418-432. doi: 10.2450/BloodTransfus.1026. Epub 2025 May 9. PMID 40423585
- See also: REDS-IV-P public website — http://redsivp.com